CLINICAL TRIAL: NCT04055311
Title: Recovery Support for Bladder Cancer Patients and Caregivers: A Multimodal Approach
Brief Title: Recovery Support for Bladder Cancer Patients and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Fox Chase Cancer Center (Other)
Responsible Party: Principal Investigator, Michael Diefenbach, Professor, Director of Behavioral Research, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 18-0400
Record Dates: First submitted 2019-07-22; First posted 2019-08-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Bladder Cancer; Patient Engagement; Patient Empowerment; Ileal Conduit
Keywords: patient focused intervention; caregiver; Internet based information; recovery support; bladder cancer; urinary diversion; neobladder
MeSH Terms: conditions — Urinary Bladder Neoplasms; Patient Participation

STUDY DESIGN:
Intervention Model Description: The RSBC intervention will be evaluated in a 12-month randomized controlled trial among patients and caregiver dyads (N=287 initial; 238 final sample) against a time and attention comparison condition that focuses on general wellness.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Participants will be randomized based on a randomization table developed by study statistician. Care providers are not informed of the assigned study condition. Patients complete assessments through Redcap survey. Data analyst will be blinded to the nature of the numerical assignment of intervention vs control condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care enhanced (Active Comparator): Bladder cancer patients & caregivers receive standard instructions about post-op care from nursing staff plus the NCI published Facing forward cancer survivorship manual.
  Interventions: Behavioral: Usual Care Enhanced
- Intervention (Experimental): Bladder cancer patients & caregivers receive standard instructions about post-op care from nursing staff plus access to Internet based software program, specifically designed for this research study. Software program contains relevant bladder cancer care instructions through videos, text, and graphics.
  Interventions: Behavioral: Cancer Resource Information Support (CRIS)

INTERVENTIONS:
Behavioral: Cancer Resource Information Support (CRIS) — Intervention support is patient initiated and accessed as needed
  Arms: Intervention
Behavioral: Usual Care Enhanced — Usual care is enhanced with the addition of the NCI Facing Forward brochure
  Arms: Usual care enhanced

SUMMARY:
For patients with certain types of bladder cancer, the removal of the bladder and the construction of an artificial bladder or reservoir are the only treatment options. Both before and after treatment, patients and caregivers face profound challenges preparing for surgery and planning for tasks during their recovery. To aid in recovery and enhance quality of life this program of research will develop and evaluate a multi-stage intervention geared towards patients and their caregivers. Part 1 of this program will have a nurse or trained health professional prepare both patients and their caregivers before treatment about the upcoming surgery. During this time the nurse will also demonstrate the necessary tools and techniques for stoma care. In addition, patients and their caregivers will receive access to a recovery website, specifically designed for bladder cancer patients to be used as a resource for after treatment. The website will be part 2 of this research and will contain important recovery information, videos about post-surgical care, testimonials by other patients and physicians and a variety of other resources. Patients and caregivers in the control group will receive the Facing Forward brochures from the National Cancer Institute in part 2. This research has been funded by the National Cancer Institute and will be the first study to address the needs of bladder cancer patients and their caregivers. The ultimate goal of the study is to reduce infections and unplanned nurse/ER visits and improve quality of life for both patients and their caregivers. This new program will be evaluated over the course of 12-months and if found successful, has the potential to be disseminated throughout the health care systems of the two study sites.

DETAILED DESCRIPTION:
Treatment for certain types of bladder cancer (BC) involves the removal of the bladder and construction of a new voiding system and is physically and psychologically profoundly challenging for patients and caregivers. Based on investigators' published literature and extensive pilot data, patients and caregivers have extensive unmet informational, social, psychological, instrumental, and medical needs from the time of diagnosis, through treatment and recovery which are not adequately addressed by health care professionals. Investigators propose to address these unmet needs through the refinement and evaluation of a comprehensive, 2-part (in-person and web-based) intervention, geared towards the patient and caregiver. Specifically, during Aim 1, the formative phase, investigators propose to further refine the newly developed intervention components with the help of an established patient/caregiver advisory board. The intervention, Recovery Support for Bladder Cancer (RSBC), consists of a pre-treatment, in-person preparatory instructional session with a trained health care professional (Module 1) to equip patients and caregivers with the skills to adjust to the upcoming treatment and recovery period. This is followed by a post-treatment, interactive web-based program (Module 2) to provide further support for both patients and caregivers to enhance quality of life (QOL) and reduce infections and nurse/ER visits. The RSBC intervention will be evaluated in a 12-month randomized controlled trial (Aim 2) among patients and caregiver dyads (N=287 initial; 238 final sample) against a time and attention comparison condition (the Facing Forward brochures). Primary outcomes for both patients and caregivers will be improved QOL, which is hypothesized to be significantly higher among participants randomized into RSBC. Secondary outcomes will be fewer infections and nurse-ER visits for patients randomized into RSBC. Aim 3 proposes moderator (i.e., age, gender, surgical diversion type) and mediator (i.e., patient activation, distress) analyses of intervention efficacy. Investigators hypothesize that RSBC will be significantly more successful among (a) older, (b) female participants, and (c) patients with a conduit diversion type. Elevated levels of patient activation (i.e., higher self-care knowledge, self-efficacy, lower distress) will mediate the intervention effects. Exploratory Aim 4 will examine the costs and potential savings associated with developing and implementing the RSBC intervention. Investigators hypothesize that initial development and implementation costs of RSBC will be offset by reduced nurse/ER visits. The scientific premise is strong and supported by an established theoretical framework, extensive pilot data and a rigorous application of clinical research methods. The proposed study is highly innovative, as it comprehensively addresses unmet needs of both patients and caregivers from pre- and (immediate) post-treatment to recovery. This is achieved through an innovative combination of in-person preparation and skill-building and web-based technology. If successful, RSBC has the potential to significantly change clinical care for patients and caregivers with BC.

ELIGIBILITY:
Inclusion Criteria:

* (a) male or female patients diagnosed with BC
* (b) undergoing bladder removal surgery and one of the following urinary diversions: 1) ileal conduit, 2) neobladder or 3) Indiana pouch.
* (c) did not need or completed neo-adjuvant chemotherapy,
* (d) able to communicate with ease in English

Exclusion Criteria:

* (a) the caregiving relationship is temporary (e.g., an out-of-town relative provides temporary support) as stated by both patient and caregiver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Quality of Life Patient: The Functional Assessment of Cancer Therapy-Bladder Cancer-Cystectomy | Baseline,
  The Functional Assessment of Cancer Therapy-Bladder Cancer-Cystectomy
Quality of Life Patient: The Functional Assessment of Cancer Therapy-Bladder Cancer-Cystectomy | 1 month
  The Functional Assessment of Cancer Therapy-Bladder Cancer-Cystectomy
Quality of Life Patient: The Functional Assessment of Cancer Therapy-Bladder Cancer-Cystectomy | 3 months
  The Functional Assessment of Cancer Therapy-Bladder Cancer-Cystectomy
Quality of Life Patient: The Functional Assessment of Cancer Therapy-Bladder Cancer-Cystectomy | 6 months
  The Functional Assessment of Cancer Therapy-Bladder Cancer-Cystectomy
Quality of Life Patient: The Functional Assessment of Cancer Therapy-Bladder Cancer-Cystectomy | 12 months
  The Functional Assessment of Cancer Therapy-Bladder Cancer-Cystectomy
Quality of Life Caregiver: The Caregiver Quality of Life Index-C | Baseline
  The Caregiver Quality of Life Index-C
Quality of Life Caregiver: The Caregiver Quality of Life Index-C | 1 month
  The Caregiver Quality of Life Index-C
Quality of Life Caregiver: The Caregiver Quality of Life Index-C | 3 months,
  The Caregiver Quality of Life Index-C
Quality of Life Caregiver: The Caregiver Quality of Life Index-C | 6 months,
  The Caregiver Quality of Life Index-C
Quality of Life Caregiver: The Caregiver Quality of Life Index-C | 12 months,
  The Caregiver Quality of Life Index-C

SECONDARY OUTCOMES:
Infection rate (biological factor) | 1 month
  Infection rate will be assessed through self-report and verified through electronic medical chart review for each patient
Infection rate (biological factor) | 3 months
  Infection rate will be assessed through self-report and verified through electronic medical chart review for each patient
Infection rate (biological factor) | 6 months
  Infection rate will be assessed through self-report and verified through electronic medical chart review for each patient
Infection rate (biological factor) | 12 months
  Infection rate will be assessed through self-report and verified through electronic medical chart review for each patient
Visiting Nurse/ER visits | 1 month
  Nurse or ER visits will be assessed through self-report and verified through electronic medical chart review
Visiting Nurse/ER visits | 3 months
  Nurse or ER visits will be assessed through self-report and verified through electronic medical chart review
Visiting Nurse/ER visits | 6 months
  Nurse or ER visits will be assessed through self-report and verified through electronic medical chart review
Visiting Nurse/ER visits | 12 months
  Nurse or ER visits will be assessed through self-report and verified through electronic medical chart review

OTHER OUTCOMES:
Exploratory Cost Analysis | 6 months
  Costs relative to the development, implementation & maintenance of the intervention and cost of post-treatment care from the medical and billing records.
Exploratory Cost Analysis | 12 months
  Costs relative to the development, implementation & maintenance of the intervention and cost of post-treatment care from the medical and billing records.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Diefenbach, PhD, Principal Investigator — Northwell Health
Locations (2):
- United States (2):
  - Northwell Health, Manhasset, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD) will be de-identified and pooled before sharing on the Open Science Framework, along with a data dictionary and statistical analysis plan for those who wish to replicate our findings or make new discoveries, using our collected data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol, including the statistical analysis plan, informed consent form, data dictionary, and de-identified, pooled individual participant data will be made available within a year of final participant data collection. We anticipate this data to be available on the Open Science Framework platform indefinitely.
Access Criteria: De-identified, pooled IPD will be made freely available on Open Science (https://osf.io/hy63z/). If additional information is requested, access can be provisioned by emailing the PI and completing a data use agreement.